CLINICAL TRIAL: NCT01744821
Title: A Randomized Controlled Pilot Trial of Vitamin D3 Replacement of Placebo Followed by Bilateral Salpingo-Oophorectomy for Women at Increased Risk of Developing Ovarian, Fallopian, or Primary Peritoneal Cancer.
Brief Title: Vitamin D for Women at Increased Risk of Developing Ovarian, Fallopian, or Primary Peritoneal Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability to recruit study subjects
Sponsor: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STU00064898
Record Dates: First submitted 2012-11-30; First posted 2012-12-07 (Estimated); Results first posted 2015-03-23 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer
Keywords: High Risk
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm A: Vitamin D3 Group (Active Comparator): Patients will take Vitamin D3 by mouth in the weeks prior to and including the morning of surgery. If blood test done at the start of the study shows that patients have a low (< or = 30 ng/ml) Vitamin D level, patients will be given two 25,000 IU Vitamin D3 Tablets (for a total of 50,000 IU) to take once a week until surgery. If baseline Vitamin D level is >30ng/ml, patients will be given on 2,000 IU Vitamin D3 tablet to take once a day until day of surgery.
  Interventions: Dietary Supplement: Arm A: Vitamin D3 Group
- Arm B: Placebo Group (Placebo Comparator): Patients will take a placebo by mouth prior to and including the morning of surgery. If bloods tests done at the start of study show that the patients have a low (< or = 30 ng/ml) Vitamin D level, patients will be given 2 placebo tablets to take once a week until surgery. If baseline Vitamin D level is > 30 ng/ml, patients will be given on placebo tablet to take once a day until surgery.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Arm A: Vitamin D3 Group
  Arms: Arm A: Vitamin D3 Group
Dietary Supplement: Placebo
  Arms: Arm B: Placebo Group

SUMMARY:
The purpose of this research is to study Vitamin D3 replacement for patients at high risk of developing ovarian, fallopian tube, or peritoneal cancer, and see if the Vitamin D3 replacement may be able to prevent the cancer.

This study is being done because in the United States ovarian cancer is the leading cause of death among women with gynecologic cancer. Women with BRCA mutations, a personal history of breast cancer, and a family history of breast and ovarian cancer are at high risk of developing ovarian, fallopian, and primary peritoneal cancer. Novel treatments other than surgery which can decrease the risk of developing ovarian, fallopian tube, and primary peritoneal cancer are important. Vitamin D has been shown to reduce the risk of developing bladder, breast, colon, endometrial, esophageal, gallbladder, gastric, lung, pancreatic, prostate, rectal, renal, vulvar and Hodgkin and non-Hodgkin lymphoma, and it may play a role in the prevention of ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be undergoing prophylactic or therapeutic oophorectomy
* Patients must be considered to be at a high risk of developing ovarian, fallopian or primary peritoneal cancer, according to 1 or more of the following characteristics:
* Patients with a BRCA mutation including variants of uncertain significance
* Patients with Lynch syndrome
* Patients with a family history that places them at high risk of developing ovarian cancer
* Patients with a personal history of breast cancer
* Patients currently taking Vitamin D prior to registration will be eligible if serum Vitamin D levels are <60ng/ml. We believe that most of these patients will be on low replacement doses of Vitamin D3 to begin with but in order to prevent against toxicity their Vitamin D3 levels will be checked at the start of the trial.
* Patients must be women age 18 and older
* Patients who are of childbearing potential and sexually active must use contraception while on study.
* Patients must have a signed and witnessed informed consent and authorization permitting release of personal health information prior to registration on the study.

Exclusion Criteria:

* Patients who are unable to take Vitamin D3 supplementation are NOT eligible
* Patients who are unwilling or unable to undergo oophorectomy are NOT eligible
* Patients with suspicious or abnormal findings on preoperative physical exam, laboratory results, or imaging studies within 4 weeks of treatment start are NOT eligible
* Patients with a GFR <59 within 4 weeks of treatment start are NOT eligible
* Patients are NOT eligible if they exhibit any contraindications within 4 weeks of treatment start to 25 (OH) D supplement including:
* Hypercalcemia (>11.5mg/dL)
* Hypervitaminosis D
* Malabsorption syndrome
* Active gallbladder disease
* Active hepatic disease
* Hypoparathyroidism
* Leukemia
* Nephrolithiasis
* Renal failure sarcoidosis
* Renal disease (eGFR<59 ml/min/1.73m2)
* Patients currently receiving digoxin are NOT eligible
* Patients who are pregnant or breastfeeding are NOT eligible. Patients must have a negative urine pregnancy test at baseline (within 4 weeks of treatment start) to confirm eligibility

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-10; Primary Completion 2014-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - NorthShore University HealthSystem, Evanston, Illinois

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants were women at high risk for ovarian cancer and undergoing a prophylactic salpingo-oophorectomy. Subjects were recruited in the outpatient gynecologic oncology clinics of the study investigators. The study opened 6/1/12 with a goal of 80 subjects. It closed on 1/12/15 with a total of 7 subjects.
Pre-assignment Details: Baseline evaluation included physical examination, personal and family history questionnaire, and blood test including serum 25(OH)D. Based on vitamin D level, subjects were randomized to 1 of 4 groups.
Groups:
- Vitamin D 50,000 IU Weekly: If Vitamin D level is ≤ 30ng/ml at baseline, randomized to 50,000 IU p.o. weekly until surgery (levels will be rechecked every 4 weeks)
- Placebo 50,000 IU Weekly: If Vitamin D level is ≤ 30ng/ml at baseline, randomized to Placebo p.o. weekly until surgery (levels will be rechecked every 4 weeks)
- Vitamin D 2,000 IU Daily: If Vitamin D level is>30ng/ml at baseline, randomized to 2000 IU p.o. daily until surgery (levels will be rechecked every 4 week)
- Placebo 2,000 IU Daily: If Vitamin D level is>30ng/ml at baseline, randomized to Placebo p.o. daily until surgery (levels will be rechecked every 4 weeks)
Period: Overall Study
Arm/Group | Vitamin D 50,000 IU Weekly | Placebo 50,000 IU Weekly | Vitamin D 2,000 IU Daily | Placebo 2,000 IU Daily
Started | 1 | 3 | 2 | 1
Completed | 1 | 3 | 2 | 1
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: With a total of 80 patients (40 per arm), assuming a Type I error rate of 5% and a power of 80, an effect size of 0.63 may be detected between patients exposed to Vitamin D supplementation and those not exposed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D 50,000 IU Weekly | Placebo 50,000 IU Weekly | Vitamin D 2,000 IU Daily | Placebo 2,000 IU Daily | Total
Number analyzed (Participants) | 1 | 3 | 2 | 1 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 2 | 1 | 7
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 2 | 1 | 7
  Male | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 3 | 2 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: The Outcomes That Will be Measured for the Primary Objectives of This Study Will be Surrogate Endpoint Biomarkers Markers of Cancer Prevention
Description: Activation of apoptosis via immunohistochemical measurement of activation of caspase activity, as well as expression of BAX and BCL-2 The primary marker outcomes will be assessed for normality and compared between groups using a two-sample t-test or a Wilcoxon rank sum test. Other markers will be compared similarly if continuous, or by Fisher's exact test if categorical.
Time Frame: Up to 24 months
Population: We failed to accrue enough patients in order to conduct this outcome measure. We collected the specimens but were unable to analyze them given the low accrual numbers.
Arm/Group | Vitamin D 50,000 IU Weekly | Placebo 50,000 IU Weekly | Vitamin D 2,000 IU Daily | Placebo 2,000 IU Daily
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Primary Outcome: Other Surrogate Endpoint Biomarkers Markers of Cancer Prevention
Description: Decrease in cellular proliferation measured by immunohistochemistry staining with KI67
Time Frame: Up to 24 months
Population: as for outcome 1
Arm/Group | Vitamin D 50,000 IU Weekly | Placebo 50,000 IU Weekly | Vitamin D 2,000 IU Daily | Placebo 2,000 IU Daily
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Review of Standard Pathologic Evaluation With Specific Attention to Histologic Markers
Description: The outcomes that will be measured for the secondary objectives of this study will include the following:
  Review of standard pathologic evaluation with specific attention to histologic markers including serous hyperplasia, tubal atypia, and p53 signature in the ovary and fallopian tube, and examine via immunohistochemistry the effects of vitamin D supplementation on expression of the TGF-beta isoforms and CYP24
Time Frame: Up to 24 months
Population: as for outcome 1
Arm/Group | Vitamin D 50,000 IU Weekly | Placebo 50,000 IU Weekly | Vitamin D 2,000 IU Daily | Placebo 2,000 IU Daily
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Review of the Differences in the Types and Incidence of Toxicities Associated With Vitamin D3 Replacement.
Description: Differences in the types and incidence of toxicities associated with Vitamin D3 replacement, specifically hypercalcemia, with increasing levels of Vitamin D3 along with the effectiveness of Vitamin D3 supplementation on increasing serum levels of Vitamin D
Time Frame: Up to 24 months
Measure: Number; unit: participants
Arm/Group | Vitamin D 50,000 IU Weekly | Placebo 50,000 IU Weekly | Vitamin D 2,000 IU Daily | Placebo 2,000 IU Daily
Number analyzed (Participants) | 1 | 3 | 2 | 1
participants
  Fatige grade 1 | 1 | 0 | 0 | 0
  Headache grade 1 | 0 | 1 | 1 | 0
  Hypercalcemia | 0 | 0 | 0 | 0
  Loss of Appetite grade 1 | 0 | 1 | 0 | 0
  Dry Mouth grade 1 | 1 | 1 | 0 | 0
  Constipation grade 1 | 1 | 0 | 0 | 0
  Weakness grade 1 | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Vitamin D 50,000 IU Weekly | Placebo 50,000 IU Weekly | Vitamin D 2,000 IU Daily | Placebo 2,000 IU Daily
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/3 | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/3 | 2/2 | 0/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin D 50,000 IU Weekly (N=1) | Placebo 50,000 IU Weekly (N=3) | Vitamin D 2,000 IU Daily (N=2) | Placebo 2,000 IU Daily (N=1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) — Grade 1
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — Grade 1
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Grade 1
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Grade 1
Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Grade1
Loss of Appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Grade 1

LIMITATIONS AND CAVEATS:
Low accrual led to this pilot study closing early. Accrual barriers included the 4-week minimum treatment time frame and narrow eligibility criteria. Small numbers prohibit meaningful analysis. Study provides important insights to recruitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No